CLINICAL TRIAL: NCT01762878
Title: A Single-Centre, Double-Blind, Placebo Controlled Two Part Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of GSK2269557 as a Dry Powder in Healthy Subjects Who Smoke Cigarettes
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Repeat Doses of the Dry Powder Formulation of GSK2269557 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116617
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: pharmacodynamics; pharmacokinetics; healthy volunteers; Pi3K-delta; GSK2269557; safety; dry powder inhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nemiralisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- GSK2269557 100 mcg arm (Experimental): Each subject will receive 4 treatments in 4 treatment periods in Part A of the study. Subjects in this arm will be randomized to receive GSK2269557 100 mcg in one of the 4 treatment periods.
  Interventions: Drug: GSK2269557
- GSK2269557 500 mcg arm (Experimental): Each subject will undergo 4 treatments in 4 treatment periods in Part A of the study. Subjects in this arm will be randomized to receive GSK2269557 500 mcg in one of the 4 treatment periods
  Interventions: Drug: GSK2269557
- GSK2269557 3000 mcg arm (Experimental): Each subject will undergo 4 treatments in 4 treatment periods in Part A of the study. Subjects in this arm will be randomized to receive GSK2269557 3000 mcg in one of the 4 treatment periods
  Interventions: Drug: GSK2269557
- Placebo arm (Placebo Comparator): The subjects will receive single dose of placebo in each treatment period of part A and repeat doses of placebo in Part B of the study.
  Interventions: Drug: Placebo
- Part B GSK2269557 arm (Experimental): The selection of total daily doses of GSK2269557 for Part B will anticipated to be the maximum well tolerated dose selected from Part A. The subjects will receive GSK2269557 in ratio of 3:1.with placebo. If the dose selected for Part B is not well tolerated on repeat dosing the dose may be reduced during Part B or given as divided doses.
  Interventions: Drug: GSK2269557

INTERVENTIONS:
Drug: GSK2269557 — Dry powder for oral inhalation (100 and 500 mcg /blister) once daily using DIKUS device. The doses of GSK2269557 planned for Part A are: 100 mcg, 500 mcg and 3000 mcg
  Arms: GSK2269557 100 mcg arm; GSK2269557 3000 mcg arm; GSK2269557 500 mcg arm; Part B GSK2269557 arm
Drug: Placebo — Dry powder for oral inhalation once daily using DIKUS device
  Arms: Placebo arm

SUMMARY:
GSK2269557 is potent and highly selective inhaled phosphoinositides 3-kinases -delta (PI3K-delta) inhibitor being developed as an anti-inflammatory agent for the treatment of inflammatory airway diseases. GSK2269557 has already been administered as a nebulized solution in single and repeat doses to humans and has been well tolerated across the range of doses used. The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of single and repeat inhaled doses of GSK2269557 as a dry powder. This study is the first administration of dry powder GSK2269557 in humans.

Part A will consist of four treatment periods separated by at least 14 days wash out periods. In each treatment period there will be 12 subjects receiving GSK2269557 and 4 subjects receiving placebo. The doses of GSK2269557 planned for Part A are 100 micrograms (mcg), 500 mcg and 3000 mcg. Blinded safety and available pharmacokinetic (PK) data will be reviewed before each dose escalation. Part B will be a parallel group design conducted in a separate group of subjects from Part A. Nine subjects will receive repeat doses of GSK2269557 and 3 subjects will receive repeat doses of placebo for 14 days. The total daily dose will be the same as the dose that was well tolerated in Part A. The study duration, including screening and follow-up, is not expected to exceed 82 days for subjects in part A and 55 days for subjects in part B of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are current daily cigarette smokers. Must have smoked regularly in the 12-month period preceding the screening visit and have a pack history of >= 5 pack years (number of pack years = number of cigarettes per day/20 x number of years smoked
* Normal spirometry (FEV1 >= 80% of predicted) at screening.
* Single QTcF < 450 milliseconds (msec); or QTcF< 480 msec in subjects with Right Bundle Branch Block
* Currently healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac testing. A subject with a clinical abnormality or laboratory parameters outside the reference range expected for them and the population being studied may be included only if the Investigator believes that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or outcomes
* Between 18 and 50 years of age inclusive, at the time of signing the informed consent
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented hysterectomy, bilateral oophorectomy or bilateral salpingectomy or postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods f they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods.
* Body weight >= 50 kilogram (kg) and body mass index (BMI) within the range 18 to 31 kg/meter^2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

* Subjects who are unable to produce a total weight of at least 0.100 grams (g) of selected sputum at screening
* Subjects whose primary consumption of tobacco is via methods other than cigarettes (manufactured or self-rolled). Primary methods of tobacco consumption that are excluded include, but are not limited to pipes and cigars
* Urinary cotinine levels at screening < 30 nanograms (ng)/mL
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* A history of congestive heart failure, coronary insufficiency or clinically significant cardiac arrhythmia that would contraindicate the subject's participation in the study
* A positive pre-study drug/alcohol screen
* A positive test for HIV antibody
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint ( approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Unable to refrain from the use of prescription or non-prescription drugs (except simple analgesics), including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* The subject has received any type of vaccination within 4 weeks of their first dose of investigational product, or are expected to be vaccinated within 4 weeks after their last dose of investigational product
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 90 day period
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated
* Subjects who have asthma or a history of asthma (except in childhood and which has now remitted)
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids from 7 days prior to the first and subsequent doses of study medication and until collection of the last PK sample for that study period

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2013-10-21 (Actual); Study Completion 2013-10-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending doses assessed by clinical monitoring of blood pressure | up to 52 days
  Blood pressure measurement will include systolic and diastolic blood pressure measured after resting in the supine position for 5 minutes
Safety and tolerability of repeat doses assessed by clinical monitoring of blood pressure | up to 24 days
  Pulse rate measurement should be done after resting in the supine position for 5 minutes
Safety and tolerability of single ascending doses assessed by pulse rate | up to 52 days
  Pulse rate measurement should be done after resting in the supine position for 5 minutes
Safety and tolerability of repeat doses assessed by pulse rate | up to 24 days
  Pulse rate measurement should be done after resting in the supine position for 5 minutes
Safety and tolerability of single ascending doses assessed by spirometry (FEV1) | up to 52 days
  Pulmonary function test measured from forced expiratory volume in 1 second (FEV1). Pulmonary function test will be repeated until three technically acceptable measurements have been made.
Safety and tolerability of repeat doses assessed by spirometry | up to 24 days
  Pulmonary function test measured from FEV1. Pulmonary function test will be repeated until three technically acceptable measurements have been made.
Safety and tolerability of single ascending doses assessed by Electrocardiogram (ECG) | up to 52 days
  12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Bazett's formula (QTcB)/ QT duration corrected for heart rate by Fridericia's formula (QTcF) intervals. ECGs will be measured after resting in supine position for 5 minutes
Safety and tolerability of repeat doses assessed by ECG | up to 24 days
  12-lead ECGs will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QTcB/QTcF intervals. ECGs will be measured after resting in supine position for 5 minutes
Safety and tolerability of single ascending doses assessed by clinical laboratory test | up to 52 days
  Clinical laboratory test includes hematology, clinical chemistry, urinalysis and additional parameters
Safety and tolerability of repeat doses assessed by clinical laboratory test | up to 24 days
  Clinical laboratory test includes hematology, clinical chemistry, urinalysis and additional parameters
Safety and tolerability of single ascending doses assessed by number of subjects with adverse events (AEs) | up to 52 days
  AEs will be collected from the start of study treatment and until the follow-up contact
Safety and tolerability of repeat doses assessed by number of subjects with AEs | up to 24 days
  AEs will be collected from the start of study treatment and until the follow-up contact

SECONDARY OUTCOMES:
Single ascending doses plasma GSK2269557 PK assessed by AUC (0-t) and AUC (0-infinity) | 2 days of each treatment period in part A. Blood samples (2 mililiter [mL]) for plasma PK parameters will be collected on Day 1(pre-dose, 0.083, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 hrs post dose) and on Day 2 (24 hrs post dose).
  To evaluate the single ascending doses PK, area under the time-concentration curve from time zero (pre-dose) to last time of quantifiable concentration (AUC[0-t]) and AUC from zero to infinity (AUC[0-infinity]) following single ascending doses will be assessed
Repeat doses plasma GSK2269557 PK assessed by AUC (0-t) and AUC (0-infinity) | 15 days of part B. Blood samples (2 mL) for plasma PK parameters will be collected on Day 1 through Day 13 (pre-dose and 0.083 hrs post dose), on Day 14 (pre-dose, 0.083, 0.5, 0.75, 1, 2, 3, 4, 6, 8, and 12 hrs post dose), and on Day 15 (24 hrs post dose
  To evaluate the repeat doses PK, (AUC[0-t]) and (AUC[0-infinity]) following repeated doses will be assessed
Single ascending doses plasma GSK2269557 PK assessed by Cmax and Ctau | 2 days of each treatment period in part A. Blood samples (2 mL) for plasma PK parameters will be collected on Day 1(pre-dose, 0.083, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 hrs post dose) and on Day 2 (24 hrs post dose).
  To evaluate the single ascending doses PK, maximum observed concentration (Cmax) and pre-dose (trough) concentration at the end of the dosing interval (Ctau) following single ascending doses will be assessed.
Repeat doses plasma GSK2269557 PK assessed by Cmax and Ctau | 15 days of part B. Blood samples (2 mL) for plasma PK parameters will be collected on Day 1 through Day 13 (pre-dose and 0.083 hrs post dose), on Day 14 (pre-dose, 0.083, 0.5, 0.75, 1, 2, 3, 4, 6, 8, and 12 hrs post dose), and on Day 15 (24 hrs post dose
  To evaluate the repeat doses PK, Cmax and Ctau following repeated doses will be assessed
Single ascending doses plasma GSK2269557 PK assessed by Tmax and T1/2 | 2 days of each treatment period in part A. Blood samples (2 mL) for plasma PK parameters will be collected on Day 1(pre-dose, 0.083, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 12 hrs post dose) and on Day 2 (24 hrs post dose).
  To evaluate the single ascending doses PK, time to occurrence of Cmax and terminal phase half-life (T1/2) following single ascending doses will be assessed.
Repeat doses plasma GSK2269557 PK assessed by Tmax and T1/2 | 15 days of part B. Blood samples (2 mL) for plasma PK parameters will be collected on Day 1 through Day 13 (pre-dose and 0.083 hrs post dose), on Day 14 (pre-dose, 0.083, 0.5, 0.75, 1, 2, 3, 4, 6, 8, and 12 hrs post dose), and on Day 15 (24 hrs post dose
  To evaluate the repeat doses PK, Tmax and T1/2 following repeated doses will be assessed.
Steady state concentration assessed by BAL concentrations of GSK2269557 and derived ELF and cell pellet deposition after repeat doses | Day 15 of Part B
  To investigate the steady-state trough concentration of GSK2269557 in lung after repeat doses, bronchial alveolar lavage (BAL) samples collected during bronchoscopy and derived epithelial lining fluid (ELF) and BAL cell pellet will be analyzed.
BAL and plasma concentrations of urea | Day 15 of Part B
  To investigate the steady-state trough concentration of GSK2269557 after repeat doses.
Single ascending doses PD effect of GSK2269557 assessed by PIP3 in sputum cells | Up to 52 days
  Sputum samples will be collected to evaluate single ascending doses pharmacodynamic (PD) effect of GSK2269557 on biomarker Phosphatidylinositol (3,4,5)-trisphosphate (PIP3) peak area as a proportion of (PIP3 peak area + PIP2 peak area) in sputum cells
Repeat doses PD effect of GSK2269557 assessed by PIP3 in sputum cells | Up to 14 days (Part B)
  Sputum samples will be collected to evaluate repeat doses PD effect of GSK2269557 on biomarker PIP3 peak area as a proportion of (PIP3 peak area + PIP2 peak area) in sputum cells

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 116617 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116617?search=study&search_terms=116617#rs
- Available data/document: Clinical Study Report: 116617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116617 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register